CLINICAL TRIAL: NCT03912818
Title: Phase 2 Open Label Study of Durvalumab With Neoadjuvant Chemotherapy in Variant Histology Bladder Cancer
Brief Title: Durvalumab and Standard Chemotherapy Before Surgery in Treating Patients With Variant Histology Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-48062; NCI-2019-01364 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BLDR0028 (Other: OnCore)
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Bladder Adenocarcinoma; Bladder Mixed Adenocarcinoma; Bladder Squamous Cell Carcinoma; Bladder Urothelial Carcinoma; Infiltrating Bladder Urothelial Carcinoma Sarcomatoid Variant; Infiltrating Bladder Urothelial Carcinoma With Giant Cells; Infiltrating Bladder Urothelial Carcinoma With Glandular Differentiation; Infiltrating Bladder Urothelial Carcinoma With Trophoblastic Differentiation; Infiltrating Bladder Urothelial Carcinoma, Clear Cell Variant; Infiltrating Bladder Urothelial Carcinoma, Micropapillary Variant; Infiltrating Bladder Urothelial Carcinoma, Nested Variant; Infiltrating Bladder Urothelial Carcinoma, Plasmacytoid Variant
MeSH Terms: interventions — Carboplatin; Cisplatin; Cystectomy; Doxorubicin; durvalumab; Gemcitabine; Methotrexate; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort II (durvalumab, cis-gem) (Experimental): Durvalumab (MEDI4736), at 1500 mg fixed dose, administered intravenously (IV) over 60 minutes. Standard chemotherapy will be administered as an IV infusion during each of the 4 cycles. Cisplatin 70 mg/m2 on Cycle Day 2, and gemcitabine 1,000 mg/m2 on Cycle Day 1 and Day 8 in 21 day cycles (3 weeks). Patients undergo cystectomy within 6 weeks.
  Interventions: Drug: Cisplatin; Procedure: Cystectomy; Biological: Durvalumab; Drug: Gemcitabine
- Cohort III (Durvalumab, carbo-gem) (Experimental): Durvalumab (MEDI4736), at 1500 mg fixed dose, administered intravenously (IV) over 60 minutes. Standard chemotherapy will be administered as an IV infusion during each of the 4 cycles. Carboplatin: AUC 5 on Cycle Day 1 and gemcitabine 1,000 mg/m2 on Cycle Day 1 and Day 8 in 21 day cycles (3 weeks). Patients undergo cystectomy within 6 weeks.
  Interventions: Drug: Carboplatin; Procedure: Cystectomy; Biological: Durvalumab; Drug: Gemcitabine
- Cohort I (durvalumab, DD MVAC) (Experimental): Durvalumab (MEDI4736), at1500 mg fixed dose, administered intravenously (IV) over 60 minutes. Standard chemotherapy will be administered as an IV infusion during each of the 4 cycles. Dose Dense Methotrexate, Vinblastine, Doxorubicin, Cisplatin (DD MVAC), in 14 day cycles (2 weeks), Methotrexate 30 mg/m2 on Cycle Day 1, Vinblastine 3 mg/m2 on Cycle Day 2, Doxorubicin 30 mg/m2 on Cycle Day 2 and Cisplatin 70 mg/m2 on Cycle Day 2. Patients undergo cystectomy within 6 weeks.
  Interventions: Drug: Cisplatin; Procedure: Cystectomy; Drug: Doxorubicin; Biological: Durvalumab; Drug: Methotrexate; Drug: Vinblastine

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Carboplat; Carboplatino; Carbosol; Paraplatin; Paraplatine
  Arms: Cohort III (Durvalumab, carbo-gem)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Briplatin; Cis-platinum; Cismaplat; Citoplatino; Plastistil; Platinol
  Arms: Cohort I (durvalumab, DD MVAC); Cohort II (durvalumab, cis-gem)
Procedure: Cystectomy — Undergo cystectomy
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxyl Daunorubicin; Rubex
  Arms: Cohort I (durvalumab, DD MVAC)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; MEDI-4736
Drug: Gemcitabine — Given IV
  Other Names: Difluorodeoxycytidine; Gemzar
  Arms: Cohort II (durvalumab, cis-gem); Cohort III (Durvalumab, carbo-gem)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Amethopterin; Brimexate; Methotrexate Methylaminopterin; Metotrexato
  Arms: Cohort I (durvalumab, DD MVAC)
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; Vinblastine Sulfate; vincaleukoblastine, sulfate
  Arms: Cohort I (durvalumab, DD MVAC)

SUMMARY:
This phase II trial studies the side effects of durvalumab and chemotherapy before surgery in treating patients with variant histology bladder cancer. Immunotherapy with monoclonal antibodies, such as durvalumab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as methotrexate, vinblastine, doxorubicin, cisplatin, gemcitabine, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving durvalumab in addition to standard chemotherapy may lead to better outcomes in patients with variant histology bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of durvalumab in combination with chemotherapy in subjects with variant histology bladder cancer.

SECONDARY OBJECTIVES:

I. To determine the percent of subjects post-neoadjuvant chemo-immunotherapy who achieve tumor stage of pT2 N0 M0 or better (pT1 N0 or pT0) at cystectomy.

II. To assess the response rate (RR) in post-neoadjuvant chemo immunotherapy as assessed by the investigator using imaging at screening and post treatment.

III. To assess the molecular characterization of tumor tissue pre-neoadjuvant therapy and at post treatment cystectomy (for subject who have persistent disease).

IV. To determine circulating free deoxyribonucleic acid (DNA) (cfDNA) (cell free DNA) at baseline, during treatment and following post treatment cystectomy using Natera sequencing platform.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT I: Patients receive durvalumab intravenously (IV) over 60 minutes on day 1. Chemotherapeutic agents will be administered as an IV infusion according to prescribing information or treatment guidance in general use by the Investigating site. Methotrexate on day 1, vinblastine IV on day 2, doxorubicin IV on day 2, and cisplatin IV on day 2. Cycles repeat every 14 days up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo cystectomy within 6 weeks.

COHORT II: Patients receive durvalumab IV over 60 minutes on day 1. Chemotherapeutic agents will be administered as an IV infusion according to prescribing information or treatment guidance in general use by the Investigating site. Cisplatin IV over 60 minutes on day 1, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo cystectomy within 6 weeks.

COHORT III: Patients receive durvalumab IV over 60 minutes on day 1.Chemotherapeutic agents will be administered as an IV infusion according to prescribing information or treatment guidance in general use by the Investigating site. Carboplatin IV on day 1, and gemcitabine IV on days 1 and 8. Cycles repeat every 21 days up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo cystectomy within 6 weeks.

After surgery, patients are followed up at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Eastern Collaborative Oncology Group (ECOG) performance status score of 0 or 1.
* Body weight > 30 kg.
* Absolute neutrophil count (ANC) >= 1500 mm^3 (within 28 days before the first study treatment).
* Hemoglobin >= 9.0 g/dL (within 28 days before the first study treatment).
* Platelet count >= 100,000 per mm^3 (within 28 days before the first study treatment).
* Serum bilirubin =< 1.5 X upper limit of normal (ULN) (within 28 days before the first study treatment). Subjects with Gilbert's syndrome will be considered after consultation with the principal investigator (PI).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X ULN (within 28 days before the first study treatment).
* For subjects who will be treated with dose dense methotrexate, vinblastine, doxorubicin, and cisplatin (DD MVAC) or cisplatin and gemcitabine (CG), creatinine clearance >= 50 mL/min as measured based on Cockcroft-Gault glomerular filtration rate estimation (within 28 days before the first study treatment).
* For subjects who will be treated with carboplatin and gemcitabine (Carbo Gem), creatinine clearance >= 30 mL/min as measured based on Cockcroft-Gault glomerular filtration rate estimation (within 28 days before the first study treatment).
* Anticipated life expectancy of >= 12 weeks as assessed by the investigator.
* Histologically proven carcinoma of the bladder of variant urothelial carcinoma histologies which include squamous, adenocarcinoma, nested, plasmacytoid, micropapillary, glandular differentiation, lipid cell, clear cell, undifferentiated, giant cell, trophoblastic, sarcomatoid, carcinosarcoma; subjects with mixed cell types are eligible.
* Clinical T stage 2 (cT2) T4a, N0 N1, M0 disease. Clinical T stage is based on the transurethral resection of bladder tumor (TURBT) sample and imaging studies. Subjects must undergo cystoscopy and TURBT as part of screening within 30 days prior to registration.
* Abdominal/pelvic imaging by computed tomography (CT) or magnetic resonance imaging (MRI) scan; chest imaging by CT scan or x-ray (CT/positron emission tomography (PET) within 30 days prior to registration.
* Resting 12 lead electrocardiogram (ECG) documenting Fridericia's correction formula (QTcF) =< 470 ms.
* Consent to provide a formalin fixed paraffin embedded (FFPE) tissue block and 1 hematoxylin and eosin (H and E) slide (preferred) or one of the following:

  * 10 unstained slides and 1 H and E slide OR
  * Tissue block punches and 1 H and E slide, OR
  * 4 to 6 cores and 1 H and E slide.
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow up.
* For female subjects:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation induced menopause with last menses > 1 year ago, had chemotherapy induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Exclusion Criteria:

* Prior treatment with systemic cytotoxic chemotherapy for muscle invasive bladder cancer (MIBC).
* Class III or IV heart failure, according to New York Heart Association Classifications. For patient on the dd MVAC or Cis-Gem arm, left ventricular ejection fraction of less than 50%
* Administration of an investigational therapeutic agent within 28 days of protocol registration.
* Current participation in a trial using an investigational agent. Subjects may participate in non-interventional, observational studies.
* Prior treatment with an anti-programmed cell death 1(PD1) or anti--programmed cell death ligand 1(PDL1) inhibitor including durvalumab.
* Receiving chronic systemic steroid therapy in dosing exceeding 10 mg daily of prednisone or equivalent per day within 7 days prior to the first dose of study treatment.
* History of another malignancy within 5 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Subjects with the following are allowed on study:

  * Adequately treated non melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
* Immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) or anti emetic during chemotherapy.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease]), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc). The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects with celiac disease controlled by diet alone.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the subject to give written informed consent.
* History of active primary immunodeficiency.
* Active infection including:

  * Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice)
  * Hepatitis B (known positive hepatitis B virus (HBV) surface antigen (HBsAg) result)
  * Hepatitis C
  * Human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies).
  * Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti HBc) and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study medication. Note: subjects, if enrolled, should not receive live vaccine while receiving study medication and up to 30 days after the last dose of study medication.
* Pregnant or lactating.
* Male or female subject of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to any of the study medications or any of the study medication excipients.
* Judgment by the investigator that the subject is unsuitable to participate in the study and the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Srinivas, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patients signed informed consent; 6 were assigned to treatment
Period: Overall Study
Arm/Group | Cohort I (Durvalumab, DD MVAC) | Cohort II (Durvalumab, Cis-gem) | Cohort III (Durvalumab, Carbo-gem)
Started | 3 | 0 | 3
Completed | 3 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Durvalumab, DD MVAC) | Cohort III (Durvalumab, Carbo-gem) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3-5 Adverse Events
Description: Graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The safety and tolerability of durvalumab in combination with chemotherapy in subjects with variant histology bladder cancer who initiate study treatment will be assessed as the number, by treatment cohort, of grade 3, 4, or 5 adverse events, considered probably or definitely related by the investigator.
Time Frame: At 120 days
Measure: Number; unit: events
Arm/Group | Cohort I (Durvalumab, DD MVAC) | Cohort III (Durvalumab, Carbo-gem)
Number analyzed (Participants) | 3 | 3
events
  Grade 3 | 1 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

2. Secondary Outcome: Proportion of Subjects Who Initiate Study Treatment and Achieve Tumor Stage of pT2 N0 M0 or Better (e.g., pT0, pT1 N0) at Cystectomy
Description: Achievement of tumor staging will be determined by pathologist at cystectomy and reported by treatment cohort. Assessed per National Comprehensive Cancer Network bladder cancer guidelines.
  * T0 N0 M0 = No evidence of primary tumor
  * T1 N0 M0 = Tumor staging by pathological assessment detected in lamina propria (T0), with no tumor positive nodes (N0).
  * T2 N0 M0 = Tumor staging by pathological assessment detected in muscularis propria (pT2), with no tumor positive nodes (N0) or tumor metastases (M0) observed.
Time Frame: At 20 weeks
Population: Participants who underwent renal cystectomy are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Durvalumab, DD MVAC) | Cohort III (Durvalumab, Carbo-gem)
Number analyzed (Participants) | 3 | 2
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Time of Consent to end of study treatment plus 90 days (average approximately 20 weeks)
Arm/Group | Cohort I (Durvalumab, DD MVAC) | Cohort III (Durvalumab, Carbo-gem)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (Durvalumab, DD MVAC) (N=3) | Cohort III (Durvalumab, Carbo-gem) (N=3)
Abcess (Infections and infestations) | 1 | 0 — Unrelated
Hypercapnia (Blood and lymphatic system disorders) | 1 | 0 — Unrelated
Cardiopulmonary Arrest (Cardiac disorders) | 1 | 0 — Unrelated
Anemia (Blood and lymphatic system disorders) | 1 | 1 — Possibly Related
Ureteral Obstruction with increased creatinine (Renal and urinary disorders) | 1 | 0 — Possibly Related
Anemia (Blood and lymphatic system disorders) | 0 | 1 — Related
Small Intestine Anastomotic Leak (Surgical and medical procedures) | 0 | 1 — Unrelated
Ureteric Anastomotic Leak (Surgical and medical procedures) | 0 | 1 — Unrelated
Sepsis (Blood and lymphatic system disorders) | 0 | 1 — Unrelated
Heart Failure (Cardiac disorders) | 0 | 1 — Possibly Related
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 — Unrelated
Dehydration (General disorders) | 0 | 1 — Related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (Durvalumab, DD MVAC) (N=3) | Cohort III (Durvalumab, Carbo-gem) (N=3)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 — Related
Anemia (Blood and lymphatic system disorders) | 1 | 1 — Related
Anorexia (Psychiatric disorders) | 1 | 0 — Related
Constipation (Gastrointestinal disorders) | 0 | 1 — Related
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Related
Dyspnea (Renal and urinary disorders) | 1 | 0 — Related
Fatigue (General disorders) | 3 | 1 — Related
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0 — Related
Hypomagnesemia (Investigations) | 0 | 1 — Related
Nausea (Gastrointestinal disorders) | 0 | 2 — Related
Paresthesia (Skin and subcutaneous tissue disorders) | 0 | 1 — Related
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 — Related
Urinary Tract Infection Not Related (Renal and urinary disorders) | 0 | 1 — Related
Watering Eyes (Eye disorders) | 0 | 1 — Related
Weight Loss (Investigations) | 0 | 1 — Related
Wound Infections (Infections and infestations) | 1 | 0 — Related
Anemia (Blood and lymphatic system disorders) | 2 | 1 — Unrelated
Creatinine Increased (Investigations) | 0 | 1 — Unrelated
Constipation (Gastrointestinal disorders) | 1 | 0 — Unrelated
Hypocalcemia (Investigations) | 0 | 1 — Unrelated
Infection around L nephrostomy tube (Renal and urinary disorders) | 1 | 0 — Unrelated
Tinnitus (Ear and labyrinth disorders) | 0 | 1 — Unrelated
Urinary Frequency (Renal and urinary disorders) | 1 | 0 — Unrelated
Weight Loss (Investigations) | 1 | 0 — Unrelated
Disequilibrium (Nervous system disorders) | 0 | 1 — Unrelated

LIMITATIONS AND CAVEATS:
The study did not achieve its planned enrollment size and did not achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT03912818/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03912818/ICF_002.pdf